CLINICAL TRIAL: NCT07077252
Title: An Open Multi-center Phase I/II Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of SCTB39G in Adult Patients With Advanced Malignant Solid Tumours
Brief Title: Phase I/II Study of SCTB39G in Advanced Solid Tumours
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sinocelltech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCTB39G-X201
Record Dates: First submitted 2025-07-11; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Advanced Malignant Solid Tumor
Keywords: Phase I/ II Study of SCTB39G in Advanced Solid Tumours

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SCTB39G (Experimental): SCTB39G of different doses, IV
  Interventions: Drug: SCTB39G

INTERVENTIONS:
Drug: SCTB39G — SCTB39G,IV

SUMMARY:
This study aims to evaluate the safety, tolerability, PK characteristics, immunogenicity, and preliminary anti-tumor efficacy of SCTB39G as a monotherapy in adult patients with advanced malignant solid tumours. This study is an open label, multicentre, dose-escalation and dose-expansion Phase I/II clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* 1.Voluntarily sign the informed consent form (ICF);
* 2.Male or female, ≥ 18 years and ≤ 70 years old;
* 3.Survival duration more than 3 months;
* 4.ECOG score ≤ 1 point;
* 5.histologically or cytologically confirmed diagnosis of advanced malignant solid tumour；
* 6.At least one measurable tumor lession according to RECIST v1.1;
* 7.Adequate organ and bone marrow function.

Exclusion Criteria:

* 1.Has participated in another clinical study within 4 weeks prior to the first dose;
* 2.Other malignancies diagnosed within 1 years prior to the enrollment;
* 3. Participants with brainstem, meningeal, spinal metastases, or compression; active central nervous system metastases;
* 4.NSCLC at high risk of bleeding; Obvious invasion of tumor into adjacent organs of esophageal lesions leads to high risk of bleeding or fistula,or participants after endotracheal stent implantation;
* 5.Participants with portal hypertension due to portal vein tumor thrombus at risk of bleeding;
* 6.Presence of pleural effusion, peritoneal effusion, or ascites;
* 7.Received chemotherapy, immunotherapy, biologic therapy, or other antitumor treatments within 4 weeks before enrollment
* 8.History of permanent discontinuation of immunotherapy due to immune-related toxicity or occurrence of ≥ Grade 3 irAEs;
* 9.Presence of any active autoimmune disease or a history of autoimmune disease with an expected recurrence;
* 10.History of severe allergies, severe drug allergies (including unapproved investigational drugs);
* 11.History of organ transplantation or stem cell transplantation;
* 12.Need for immunosuppressive drugs within 2 weeks prior to enrollment or anticipated during the study;
* 13.Pregnant or breastfeeding female.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-28 (Estimated); Primary Completion 2027-09-26 (Estimated); Study Completion 2027-10-17 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting toxicity(DLT) | From Day 0 up to Day 21
  Incidence of dose-limiting toxicities up to the Day 21 visit
Objective response rate (ORR) | Up to 2 years
  The ORR is defined as the proportion of subjects with confirmed CR or confirmed PR, based on RECIST Version 1.1

SECONDARY OUTCOMES:
Disease control rate (DCR) | Up to 2 years
  The DCR is defined as the proportion of subjects with CR, PR, or SD based on RECIST Version 1.1.
Progression-free survival (PFS) | Up to 2 years
  Progression-free survival is defined as the time from the start of treatment with SCTB39G until the first documentation of disease progression or death due to any cause, whichever occurs first.
Overall survival (OS) | Up to 2 years
  Overall survival is defined as the time from the start of treatment with SCTB39G until death due to any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No